CLINICAL TRIAL: NCT02092753
Title: Ketogenic Or LOGI Diet In a Breast Cancer Rehabilitation Intervention (KOLIBRI)
Acronym: KOLIBRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Marc Sütterlin, MD, PhD, MD, Universitätsmedizin Mannheim
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: KOLIBRI
Record Dates: First submitted 2014-02-26; First posted 2014-03-20 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Quality of Life
Keywords: Ketogenic diet, logi diet, breast cancer, rehabilitation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard diet (Placebo Comparator): Standard diet (SD): Nutrition following the standard recommendations of the German society for nutrition
  Interventions: Other: Standard diet (SD)
- Ketogenic diet (Experimental): Nutritional intervention: Ketogenic diet (KD).
  Intervention: Nutritional support (hospital) + self support (outpatient phase) with KD
  Interventions: Other: Experimental 1: Ketogenic diet (KD).
- Logi diet (Experimental): Nutritional intervention: low glycämic and insulinemic" diet (LOGI)
  Intervention: Nutritional support (hospital) + self support (outpatient phase) with LOGI
  Interventions: Other: Experimental 2: "Low glycämic and insulinemic" diet (LOGI)

INTERVENTIONS:
Other: Standard diet (SD) — Nutrition intervention following the recommendations of the germans society for nutrition (DGE)
  Arms: Standard diet
Other: Experimental 1: Ketogenic diet (KD). — Nutritional intervention: recommendations to follow a ketogenic diet
  Arms: Ketogenic diet
Other: Experimental 2: "Low glycämic and insulinemic" diet (LOGI) — Nutritional intervention: patients were instructed to follow the "LOGI" diet regimen
  Arms: Logi diet

SUMMARY:
The aim of the study is to analyze if a ketogenic diet (KD) compared to either a "low glycämic and insulinemic" (LOGI) diet or to a standard diet (SD) is feasible, safe and tolerable and will improve quality of life and physical performance in patients with Breast Cancer during the rehabilitation phase.

It will be an open-label trial of nutritional intervention for 20 weeks spanning three phases: 3 weeks of stationary intervention, 16 weeks of outhouse phase and one final week of stationary intervention.

DETAILED DESCRIPTION:
Cancer patient's whole body metabolism is characterized by an increased fat oxidation rate and a decrease ability to metabolize glucose for energy demands (insulin resistance). In preliminary studies it was shown, that a fat rich diet allows to spare muscle mass from being reduced due to catabolic mechanisms. The resulting better body composition relates to less fatigue and higher quality of life, the latter was shown in advanced cancer patients for a ketogenic diet.

The aim of the KOLIBRI-study is to analyze if a very fat rich ketogenic diet (KD) or a moderate fat rich "low glycämic and insulinemic" (LOGI) diet compared to a standard low fat diet (SD) are feasible, safe and tolerable and will improve quality of life and physical performance in patients with Breast Cancer during the rehabilitation phase.

The most stringent nutritional regime high in fat and low in carbohydrates is the ketogenic diet (KD) comprised of at least 75% of daily calories via fat (derived from several plant oils, nuts, avocado, butter, cream, cheese, eggs, fatty fish and fat rich meat), balanced in protein (1.4 g/kg body weight/day) and very low in carbohydrates (approx. 20-30 grams per day, derived from salad, vegetable, some berries or fruits, and milk products like yoghurt).

A less strict but even lower in carbohydrates and richer in fat and protein than a standard diet is the LOGI regimen. It allows up to 120 grams of carbohydrates (inclusion of more vegetable and fruit and rare grains and potatoes compared to KD), is high in protein (1.7 g/kg body weight/day) and rich in fat (remaining calories) The control nutritional regime follows the standard recommendations of the German society for nutrition (DGE) and is comprised of at least 50% of the daily energy derived from carbohydrates, 0.8 grams/kg of body weight protein and 30% of daily energy expenditure from fat.

It will be an open-label trial of nutritional intervention for 20 weeks spanning three phases:

The first phase spans 3 weeks of stationary intervention in a hospital (location: Bad Kissingen, Bavaria, Germany) with the initial examination (medical, body composition, food preferences, quality of life, blood samples, physical performance) followed by implementation of the allocated diet and respective training of the patients in diet calculation, cooking and realization of the diet regimen in routine daily life.

The second phase encompasses16 weeks of an outhouse phase with continuing the selected nutritional regime under close contact and supervision of the study team accompanied by urine measurements (KD group), food diaries, questionnaires covering the quality of life and one blood sample) The third phase of the study represents one week of stationary intervention at the hospital with the final examination and further teaching in eiterh sticking to the selected diet or in changing the diet to the individually preferred one.

ELIGIBILITY:
Inclusion Criteria:

1. Consenting women aged 18 - 70 years.
2. Primary or recurrent breast cancer after primary standard therapy during the standard rehabilitation phase
3. Karnofsky Index >70.
4. Willing and being able to follow the allocated dietary regime for 20 weeks

Exclusion Criteria:

1. Patients with additional malignant tumors at the time of the recruitment
2. Participation at other trials
3. Dementia or other clinically relevant alterations of the mental status which could impair the ability of the patient to apply to the diet or understand the informed consent of the study
4. Not able to follow the teaching due to deficits in teaching language (German)
5. Metabolic aberration banning fat rich nutrition or were a KD is contraindicated
6. Expected life span < 12 month
7. Insulin dependent Diabetes
8. Decompensated heart failure (NYHA > 2)
9. Myocardial infarction within the last 6 months, symptomatic atrial fibrillation
10. Severe acute infection
11. Pregnancy
12. Pancreatic insufficiency

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2014-03; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Quality of life | It will be an open-label trial of nutritional intervention for 20 weeks spanning three phases: 3 weeks of stationary intervention, 16 weeks of outhouse phase and one final week of stationary intervention.
  To study the effect of a ketogenic diet (KD) or a low glycämic and insulinemic diet (LOGI) compared to a standard diet (SD) on quality of life in patients with Breast Cancer during the rehabilitation phase.
  This will be done by comparing the results of the EORTC QLQ-30 and the QLQ-BR23 questionnaires.

SECONDARY OUTCOMES:
Safety | see below (description)
  For all patients in the three groups (KD, LOGI and SD ) in parallel:
  Feasibility measured as average calorie and carbohydrate intake per day during weeks 1-20 as documented by food diary at one random day/week Safety as defined as number of patients with adverse events [ Time Frame: weeks 1-20] Ketosis as dokumented daily in urine and blood [Time Frame: days 1-21] and in urine daily [Time Frame: week 4-20) Physical performance as obtained by spiroergometry [Time frame: day 1, day 21 and week 20] Body composition as analyzed by standard-Bioimpedance analysis(BIA), Dual- measurement [Time frame: day 1, 21 and week 20] Metabolic parameters (triglycerides, cholesterine, glucose, insulin, IGF-1) in patients serum via standard laboratory procedure [Time frame: day 1, 21, week 11 and 20]
Tolerability | see below
  For all patients in the three groups (KD, LOGI and SD ) in parallel:
  Feasibility measured as average calorie and carbohydrate intake per day during weeks 1-20 as documented by food diary at one random day/week tolerability as defined as number of patients with adverse events [ Time Frame: weeks 1-20] Ketosis as dokumented daily in urine and blood [Time Frame: days 1-21] and in urine daily [Time Frame: week 4-20) Physical performance as obtained by spiroergometry [Time frame: day 1, day 21 and week 20] Body composition as analyzed by standard-Bioimpedance analysis(BIA), Dual- measurement [Time frame: day 1, 21 and week 20] Metabolic parameters (triglycerides, cholesterine, glucose, insulin, IGF-1) in patients serum via standard laboratory procedure [Time frame: day 1, 21, week 11 and 20]

CONTACTS AND LOCATIONS:
Overall Officials: Marc Sütterlin, MD, Prof., Study Chair — Department of Obstetrics and Gynecology, University Hospital Mannheim, University of Heidelberg, Mannheim, Germany; Monika Reuss-Borst, MD, Prof., Study Director — Rehaklinik Am Kurpark, Bad Kissingen, Germany
Locations (1):
- Rehaklinik Am Kurpark, Bad Kissingen, Baden-Wurttemberg, Germany

REFERENCES:
- [Background] Woolf EC, Scheck AC. The ketogenic diet for the treatment of malignant glioma. J Lipid Res. 2015 Jan;56(1):5-10. doi: 10.1194/jlr.R046797. Epub 2014 Feb 6. PMID 24503133
- [Background] Klement RJ, Frobel T, Albers T, Fikenzer S, Prinzhausen J, Kämmerer U. A pilot case study on the impact of a self-prescribed ketogenic diet on biochemical parameters and running performance in healthy and physically active individuals. NuMe 2013; 1(1):1-32
- [Background] Fine EJ, Segal-Isaacson CJ, Feinman RD, Herszkopf S, Romano MC, Tomuta N, Bontempo AF, Negassa A, Sparano JA. Targeting insulin inhibition as a metabolic therapy in advanced cancer: a pilot safety and feasibility dietary trial in 10 patients. Nutrition. 2012 Oct;28(10):1028-35. doi: 10.1016/j.nut.2012.05.001. Epub 2012 Jul 26. PMID 22840388
- [Background] Kossoff EH, Hartman AL. Ketogenic diets: new advances for metabolism-based therapies. Curr Opin Neurol. 2012 Apr;25(2):173-8. doi: 10.1097/WCO.0b013e3283515e4a. PMID 22322415
- [Background] Klement RJ, Kammerer U. Is there a role for carbohydrate restriction in the treatment and prevention of cancer? Nutr Metab (Lond). 2011 Oct 26;8:75. doi: 10.1186/1743-7075-8-75. PMID 22029671
- [Background] Seyfried TN, Marsh J, Shelton LM, Huysentruyt LC, Mukherjee P. Is the restricted ketogenic diet a viable alternative to the standard of care for managing malignant brain cancer? Epilepsy Res. 2012 Jul;100(3):310-26. doi: 10.1016/j.eplepsyres.2011.06.017. Epub 2011 Aug 31. PMID 21885251
- [Background] Schmidt M, Pfetzer N, Schwab M, Strauss I, Kammerer U. Effects of a ketogenic diet on the quality of life in 16 patients with advanced cancer: A pilot trial. Nutr Metab (Lond). 2011 Jul 27;8(1):54. doi: 10.1186/1743-7075-8-54. PMID 21794124
- [Background] Kossoff EH, Borsage JL, Comi AM. A pilot study of the modified Atkins diet for Sturge-Weber syndrome. Epilepsy Res. 2010 Dec;92(2-3):240-3. doi: 10.1016/j.eplepsyres.2010.09.008. Epub 2010 Oct 8. PMID 20934305
- [Background] Masko EM, Thomas JA 2nd, Antonelli JA, Lloyd JC, Phillips TE, Poulton SH, Dewhirst MW, Pizzo SV, Freedland SJ. Low-carbohydrate diets and prostate cancer: how low is "low enough"? Cancer Prev Res (Phila). 2010 Sep;3(9):1124-31. doi: 10.1158/1940-6207.CAPR-10-0071. Epub 2010 Aug 17. PMID 20716631
- [Background] Seyfried BT, Kiebish M, Marsh J, Mukherjee P. Targeting energy metabolism in brain cancer through calorie restriction and the ketogenic diet. J Cancer Res Ther. 2009 Sep;5 Suppl 1:S7-15. doi: 10.4103/0973-1482.55134. PMID 20009300
- [Background] Chu-Shore CJ, Thiele EA. Tumor growth in patients with tuberous sclerosis complex on the ketogenic diet. Brain Dev. 2010 Apr;32(4):318-22. doi: 10.1016/j.braindev.2009.04.009. Epub 2009 May 13. PMID 19443154
- [Background] Kossoff EH, Turner Z, Bergey GK. Home-guided use of the ketogenic diet in a patient for more than 20 years. Pediatr Neurol. 2007 Jun;36(6):424-5. doi: 10.1016/j.pediatrneurol.2007.01.013. PMID 17560509
- See also: Hompage of the clinic in which the study is about to be accomplished. — http://www.rehaklinik-am-kurpark.de